CLINICAL TRIAL: NCT02832362
Title: A Randomized, Parallel-Group, Placebo-Controlled Study to Evaluate the Local Nasal Tolerability and Safety of 1146A in Healthy Adult Subjects
Brief Title: Local Nasal Tolerability and Safety Study of 1146A in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 205636
Record Dates: First submitted 2016-06-29; First posted 2016-07-14 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold | interventions — carbomer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Carbomer 980 (Experimental): Participants will be administered test product (nasal spray) containing 0.5% carbomer 980, 4 times per day (i.e. 3 actuations per nostril per dose; each actuation will be 140 mcL, equivalent to 140 mg).
  Interventions: Drug: Carbomer 980
- Placebo (Placebo Comparator): Participants will be administered reference product (nasal spray) containing vehicle without carbomer 980, 4 times per day (i.e. 3 actuations per nostril per dose; each actuation will be 140 mcL, equivalent to 140 mg).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Carbomer 980 — Test product containing 0.5% carbomer 980 gel
  Arms: Carbomer 980
Other: Placebo — Reference product containing vehicle without 0.5% carbomer 980 gel
  Arms: Placebo

SUMMARY:
This will be a single-center, randomized, parallel-group, placebo-controlled study to assess the local nasal tolerability and safety of multiple administrations of topically (intranasally) administered 1146A delivered by a nasal spray applicator in healthy adult participants

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form. Willing to be confined for 9 days (8 nights) and acceptance of standardized food and beverages throughout the confined study period
* Aged between 18 and 55 years inclusive
* Male or female
* Good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant and relevant abnormalities in medical history or upon physical and nasal examinations
* Participant is free of any disease or concomitant treatment that could interfere with the interpretation of the study results as determined by the investigator or the sponsor's medical officer
* Females of childbearing potential who are, in the opinion of the investigator, practicing a reliable method of contraception. Adequate contraception is defined as abstinence, oral contraceptive, either combined or progestogen alone or injectable progestogen or implants of levonorgestrel or estrogenic vaginal ring or percutaneous contraceptive patches or intrauterine device or intrauterine system or double barrier method (condom or occlusive cap [diaphragm or cervical vault caps] plus spermicidal agent [foam, gel, film, cream, suppository]) or male partner sterilization prior to the female participant's entry into the study, and this male is the sole partner for that participant

Exclusion Criteria:

* Women who have a positive urine pregnancy test
* Women who are breast-feeding
* History of malignancy or neoplastic disease of any organ system (except for localized basal cell skin carcinoma), treated or untreated, within the past 5 years prior to screening, regardless of whether there is evidence of local recurrence or metastases, clinically relevant chronic or acute infectious illnesses or febrile infections within two weeks prior to start of the study, History (within 5 years prior to study start) or any evidence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinological, metabolic, autoimmune, neurological, psychiatric or other diseases at screening, participants who have used medications or therapies that could interfere with study evaluations and have not had the proper washout period from these medications or therapies or are anticipated to require any concomitant intranasal medication during that period or at any time throughout the study, any condition that prohibits the participant from actuating nasal spray devices (severe rheumatoid arthritis; deformed hands and fingers; missing fingers), Nasal disease(s) likely to affect deposition of intranasal medication, such as acute or chronic sinusitis, rhinitis medicamentosa, clinically significant polyposis, or clinically significant nasal structural abnormalities
* Known or suspected intolerance or hypersensitivity to any of the study medications, excipients, investigational device material, or to medications of similar chemical classes, any history of drug hypersensitivity, asthma, urticaria, or other significant allergic diathesis, known or suspected contraindications, including history of allergy, or photosensitivity to study medication/s
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of screening or 5 half-lives of the other clinical studies investigational drug, whichever is longer, Previously enrolled in the current study
* Current smoker or smoked or used nicotine containing products within 5 years of screening, history (within 5 years prior to study start) or evidence of illicit drug abuse or if the investigator suspects current drug use with drug classes that include but are not limited to barbiturates, amphetamines, benzodiazepines, cocaine, opiates, cannabis or any other illicit drugs (verified by urine drug screening or other reliable evidence), history or evidence of current alcohol abuse or if participant reports a regular average alcohol consumption exceeding 18 g (women) or 35 g (men) of pure alcohol per day, i.e. 1 drink/day for women or 2 drinks/day for men (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor) within 6 months of screening
* Non-acceptance of standardized food and beverages throughout each confined study period, Ingestion of food containing poppy seeds (muffins, bagels, cakes, etc) within 24 hours of admission to the study site
* Persons directly or indirectly involved in the execution of this protocol, including employees of the contract research organization (CRO) and persons related to them, an employee of the sponsor or the study site or members of their immediate family
* On nasal examination, the presence of any superficial or moderate nasal mucosal erosion, nasal mucosal ulceration, or nasal septum perforation (Grade 1B - 4) during the screening visit or Day -1, Participants with difficulty in using the nasal spray applicator, "Vulnerable" individual (as defined by the Institutional Review Board (IRB) e.g. incarcerated person), any condition not identified in the protocol that in the opinion of the investigator would confound the evaluation and interpretation of the study data or may put the participant at risk, no consumption of alcohol-containing products within 24 hours before confinement and throughout confined study period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-11 (Actual); Primary Completion 2016-07-10 (Actual); Study Completion 2016-07-18 (Actual)

PRIMARY OUTCOMES:
Incidences of nasal mucosal changes of ≥ Grade 1B | Baseline to Day 8
  The investigators will perform a thorough examination using nasal mucosal grading scale: Grade 0 = No abnormal findings, Grade 1A = focal nasal mucosal irritation (inflammation, erythema or hyperemia), Grade 1B = superficial nasal mucosal erosion, Grade 2 = moderate nasal mucosal erosion
Incidence of moderate or severe mucosal bleeding | Baseline to Day 8
  The investigators will perform a thorough examination using mucosal bleeding scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe
Incidence of moderate or severe crusting of mucosa | Baseline to Day 8
  The investigators will perform a thorough examination using crusting of mucosa scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe

SECONDARY OUTCOMES:
Adverse events | Baseline to Day 8
  All adverse events reported by participants will be recorded.
Change from baseline in Blood pressure | Baseline to Day 8
  Systolic and diastolic BP will be measured three times after the participant has been sitting for 5 minutes using an automated validated device, e.g. OMRON, with an appropriately sized cuff. The repeat sitting measurements will be made at 1-2 minute intervals and the mean/average of the three measurements will be recorded.
Change from baseline in pulse | Baseline to Day 8
  Pulse will be measured three times after the participant has been sitting for 5 minutes using an automated validated device, e.g. OMRON, with an appropriately sized cuff. The repeat sitting measurements will be made at 1-2 minute intervals and the mean/average of the three measurements will be recorded.
Change from baseline in respiration rate | Baseline to Day 8
  The rate will be measured by counting the number of breaths for one minute (counting how many times the chest rises).
Change from baseline in oral body temperature | Baseline to Day 8
  Oral body temperature will be measured. Reference range (Oral body temperature between 35.0 º Celsius (C) and 37.5 ºC)
Change from baseline in Hematology | Baseline to Day 8
  Hemoglobin (Hb), hematocrit (Ht), red blood cell (RBC) count (including mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), mean corpuscular hemoglobin concentration (MCHC), white blood cell (WBC) count with differential and platelet count will be measured.
Change from baseline in clinical Chemistry | Baseline to Day 8
  Electrolytes (sodium, potassium, chloride, calcium, phosphorous), substrates (Blood Urea Nitrogen [BUN], creatinine, total bilirubin, total protein, albumin, uric acid, and C-reactive protein), and enzymes (aspartate amino transferase [AST], alanine amino transferase [ALT], alkaline phosphatase (ALP), gamma glutamyl transferase [GGT], creatine kinase [CK]) will be measured.
Change from baseline in virus Serology | Baseline to Day 8
  Serology will be performed only for Hepatitis B Surface Antigen (HBs Ag), Hepatitis B core antibody [anti-HBc] (Immunoglobulin G [IgG] + Immunoglobulin M [IgM]), anti-HCV Ab [Hepatitis C Virus antibody], Human Immunodeficiency Virus [HIV] 1 and HIV 2 antibodies.
Change from baseline in urinalysis | Baseline to Day 8
  Specific gravity, nitrite, protein including microalbuminuria, glucose, ketones as well as blood WBC and RBC sediments will be assessed. (
Change from baseline in urine drug & cotinine screen | Baseline to Day 8
  : Urine will be collected and tested for cotinine and the following drugs or illicit substances: barbiturates, benzodiazepines, amphetamines, cocaine, opiates, and cannabis.
Change from baseline in pregnancy and assessments of fertility | Baseline to Day 8
  A urine dipsick test will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Québec, Quebec, Canada

REFERENCES:
- See also: Results for Study 205636 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/205636?search=study&study_ids=205636#rs